CLINICAL TRIAL: NCT07279662
Title: Comparative Study on the Effects of Conventional and Skeletal Anchorage Supported Face Mask Applications on Dentofacial Structures Following the Alt-RAMEC Protocol
Brief Title: Comparison of Skeletal Anchorage Versus Conventional Tooth-Borne Face Mask Therapy Following the Alt-RAMEC Protocol
Acronym: MiniFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murat Kaan Erdem (Other)
Responsible Party: Sponsor-Investigator, Murat Kaan Erdem, PhD, DDS, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUDHF-FM-ALT-RAMEC-2025
Record Dates: First submitted 2025-11-28; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Class III Malocclusion; Skeletal Malocclusion; Maxillary Deficiency
Keywords: Face Mask Therapy; Growing Patients; Cephalometric Evaluation; Class III Orthodontic Treatment; Maxillary Protraction; Alt-RAMEC Protocol; Zygomatic Buttress Miniscrew; Miniscrew Anchorage; Skeletal Anchorage
MeSH Terms: conditions — Malocclusion, Angle Class III; Retrognathia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel treatment groups: skeletal anchorage-supported face mask therapy or conventional tooth-borne face mask therapy.
Masking Description: Treatment providers and participants could not be masked due to the nature of orthodontic appliances.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skeletal Anchorage Face Mask Group (Miniscrew/FM) (Experimental): Participants underwent the Alternate Rapid Maxillary Expansion and Constriction (Alt-RAMEC) protocol followed by maxillary protraction using skeletal anchorage. Two 2×11 mm miniscrews were placed in the zygomatic buttress region to directly apply orthopedic force to the maxilla. Face mask elastics delivering approximately 400 g of bilateral force at a 30° downward angle to the occlusal plane were worn 18-20 hours per day until a positive overjet was achieved.
  Interventions: Device: Tooth-Borne Maxillary Protraction Appliance
- Conventional Face Mask Group (Appliance/FM) (Active Comparator): Participants underwent the Alternate Rapid Maxillary Expansion and Constriction (Alt-RAMEC) protocol followed by maxillary protraction using a tooth-borne Hyrax expansion appliance with hooks for force application. Face mask elastics delivering approximately 400 g of bilateral force at a 30° downward angle to the occlusal plane were worn 18-20 hours per day until a positive overjet was achieved.
  Interventions: Device: Skeletal Anchorage Supported Maxillary Protraction

INTERVENTIONS:
Device: Skeletal Anchorage Supported Maxillary Protraction — Maxillary protraction using skeletal anchorage placed in the zygomatic buttress region following the Alt-RAMEC protocol. Two 2×11 mm miniscrews were inserted under local anesthesia, and protraction elastics delivering approximately 400 g of bilateral force at a 30° downward angle to the occlusal plane were attached to the face mask. Patients were instructed to wear the face mask for 18-20 hours per day until a positive overjet was achieved.
  Arms: Conventional Face Mask Group (Appliance/FM)
Device: Tooth-Borne Maxillary Protraction Appliance — Maxillary protraction performed using a Hyrax-type tooth-borne expansion appliance equipped with anterior hooks after completion of the Alt-RAMEC protocol. Face mask elastics delivering approximately 400 g of bilateral force at a 30° downward angle to the occlusal plane were attached to the appliance. Patients were instructed to wear the face mask for 18-20 hours per day until a positive overjet was achieved.
  Arms: Skeletal Anchorage Face Mask Group (Miniscrew/FM)

SUMMARY:
This study investigated two different methods of maxillary protraction in growing patients with skeletal Class III malocclusion characterized by maxillary deficiency. All participants underwent the Alternate Rapid Maxillary Expansion and Constriction (Alt-RAMEC) protocol to mobilize the circummaxillary sutures. Following this, maxillary protraction was performed using either skeletal anchorage with miniscrews placed in the zygomatic buttress region or a conventional tooth-borne rapid maxillary expansion appliance. Cephalometric radiographs were taken before treatment, after the Alt-RAMEC protocol, and after completion of face mask therapy to evaluate skeletal and dentoalveolar changes. The study aimed to determine whether skeletal anchorage provides greater maxillary advancement and reduced dental side effects compared to conventional tooth-borne anchorage.

DETAILED DESCRIPTION:
Skeletal Class III malocclusion with maxillary deficiency can negatively affect facial profile, occlusal function, and craniofacial growth. Early orthopedic intervention may help redirect growth and improve skeletal relationships. The Alternate Rapid Maxillary Expansion and Constriction (Alt-RAMEC) protocol has been introduced to enhance maxillary protraction by promoting greater disarticulation of the circummaxillary sutures.

In this prospective study, participants were randomly assigned to one of two treatment groups. Both groups used the same sequence of Alt-RAMEC activation over approximately seven weeks. In the skeletal anchorage group, miniscrews (2×11 mm) were placed in the zygomatic buttress region to directly apply orthopedic forces to the maxilla. In the conventional group, protraction forces were applied from hooks on a tooth-borne maxillary expansion appliance. In both groups, face mask therapy was performed with approximately 400 g of bilateral force applied at a 30-degree angle to the occlusal plane, worn 18-20 hours per day until a positive overjet was achieved.

Standardized lateral cephalometric radiographs were obtained at three time points: before treatment, after completion of the Alt-RAMEC protocol, and after completion of face mask therapy. Skeletal and dentoalveolar measurements were used to assess treatment effects. Primary outcomes focused on the forward movement of the maxilla, while secondary outcomes evaluated maxillary incisor inclination, molar position, mandibular rotations, and overjet correction.

This study aimed to clarify whether skeletal anchorage results in greater skeletal maxillary advancement and reduced dental compensation compared with conventional tooth-borne anchorage during facemask therapy in growing Class III patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 13 years.
* Skeletal Class III malocclusion with maxillary retrognathia (ANB < 0°).
* Normal or increased vertical growth pattern (SN-GoGn < 39°).
* Retrusive nasomaxillary region and/or upper lip.
* Good oral hygiene.
* No contraindication for orthodontic treatment.
* Written informed consent obtained from parents/guardians.

Exclusion Criteria:

* Systemic diseases or conditions affecting bone metabolism.
* Craniofacial syndromes or congenital anomalies.
* Functional Class III due to habitual occlusal interference.
* Previous orthodontic or orthopedic treatment.
* Severe mandibular prognathism without maxillary involvement.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Change in SNA Angle | From baseline to 10 months
  The SNA angle measures the sagittal position of the maxilla relative to the cranial base. An increase in this value indicates forward movement of the maxilla. The change in SNA (in degrees) will be compared within each group and between treatment groups.

SECONDARY OUTCOMES:
Change in A-Point to Vertical Reference Distance (A-Tvert.) | From baseline to 10 months
  A-Tvert. measures the sagittal position of Point A relative to a vertical craniofacial reference plane. An increase in this distance indicates forward movement of the maxilla. The change will be compared within groups and between treatment groups to assess the skeletal effect of protraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset includes identifiable cephalometric imaging and clinical information from pediatric participants.